CLINICAL TRIAL: NCT00612469
Title: Sodium Fluoride, Chlorhexidine and Vancomycin Effect in the Inhibition of Mutans Streptococci in Children With Dental Caries: a Randomized, Double-Blind Clinical Trial
Brief Title: The Use of Antimicrobial Agents in the Inhibition of Mutans Streptococci in Children With Dental Caries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal do Ceara (Other)
Responsible Party: Cristiane Sá Roriz Fonteles, Department of Clinical Dentistry, Federal University of Ceará
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 270/05
Record Dates: First submitted 2008-01-29; First posted 2008-02-11 (Estimated); Last update posted 2008-02-11 (Estimated); Status verified 2007-12

CONDITIONS: Dental Caries
Keywords: dental caries; vancomycin; chlorhexidine; sodium fluoride; mutans streptococci
MeSH Terms: conditions — Dental Caries | interventions — Sodium Fluoride; Vancomycin; chlorhexidine gluconate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- NaF (Placebo Comparator): Sodium fluoride application
  Interventions: Drug: Sodium Fluoride
- V3 (Experimental): Topical application of 3% vancomycin
  Interventions: Drug: vancomycin hydrochloride
- V10 (Experimental): Topical application of 10% vancomycin
  Interventions: Drug: vancomycin hydrochloride
- CHX (Active Comparator): Topical application of 1% chlorhexidine
  Interventions: Drug: chlorhexidine digluconate

INTERVENTIONS:
Drug: Sodium Fluoride — Topical application of 1.23% sodium fluoride to the dentition, every 24 hours, during 6 consecutive days
  Arms: NaF
Drug: vancomycin hydrochloride — Topical application of 3% vancomycin hydrochloride to the dentition, every 24 hours, during 6 consecutive days
  Other Names: Vanclomin, Laboratório Teuto Brasileiro S.A., Goiás, Brazil
  Arms: V3
Drug: vancomycin hydrochloride — Topical application of 10% vancomycin hydrochloride to the primary dentition, every 24 hours, during 6 consecutive days
  Other Names: Vanclomin, Laboratório Teuto Brasileiro S.A., Goiás, Brazil
  Arms: V10
Drug: chlorhexidine digluconate — Topical application of 1% chlorhexidine digluconate to the dentition, every 24 hours, during 6 consecutive days
  Arms: CHX

SUMMARY:
The aim of the present study was to compare salivary MS levels in four different groups of children with caries, that have been submitted to intraoral topical treatment with either 1,23% sodium fluoride, 1% chlorhexidine, 3% or 10% vancomycin, during 6 consecutive days. This clinical trial was designed to test two different hypotheses. First, that topical vancomycin would be more effective than chlorhexidine and sodium fluoride in salivary MS reduction. Secondly, a 6-day antimicrobial treatment with either one of these agents would produce a long lasting MS suppression, dispensing repeated antibacterial treatments.

DETAILED DESCRIPTION:
The present study aimed to compare the effect of sodium fluoride, chlorhexidine and vancomycin on salivary mutans streptococci (MS) levels, on a double-blind, randomized clinical trial. Sixty-nine healthy volunteers, aged 4-8 years, with at least one active carious lesion and no previous history of allergies were selected to participate in the study. A gel formulation containing 1.23% sodium fluoride, 1% chlorhexidine, 3% or 10% vancomycin was topically administered to the dentition every 24 hours, during 6 consecutive days. Salivary MS levels were measured at baseline (D1), on the 6th (D6), 15th (D15) and 30th day (D30). For microbiological analysis, MSB agar medium was used.

ELIGIBILITY:
Inclusion Criteria:

* Generally healthy children
* Children with at least one carious cavitated or non-cavitated lesion
* Must be able to spit
* Must be able to collaborate during clinical intervention

Exclusion Criteria:

* Children with history of allergies or allergic diseases, e.g. asthma, urticaria, rhinitis, sinusitis, or intra-oral soft tissue lesions
* Children who underwent antibiotic treatment during the course of this clinical trial
* Children with developmental disabilities
* Children with no clinical signs dental caries

Ages: 4 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 69 (Actual)
Dates: Start 2005-10; Primary Completion 2006-07 (Actual); Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
Salivary mutans streptococci levels prior to treatment, on the last day of treatment (day 6), two weeks after day 1 and 30 days after day 1. | 30-day observational period for each subject

SECONDARY OUTCOMES:
Number of new carious lesions within the different study groups 12 months after treatment discontinuation. | one year

CONTACTS AND LOCATIONS:
Overall Officials: Cristiane SR Fonteles, DDS, MS, PhD, Principal Investigator — Federal University of Ceará
Locations (1):
- School of Dentistry, Department of Clinical Dentistry, Federal University of Ceara, Fortaleza, Ceará, Brazil